CLINICAL TRIAL: NCT02129140
Title: Observational Study to Evaluate Single-Staged Open Complex Ventral Incisional Hernia Repair Using a Biologic Mesh (Cook Biodesign) for Midline Fascial Closure Reinforcement
Brief Title: Observational Study to Evaluate Ventral Incisional Hernia Repair Using a Biologic Mesh (Cook Biodesign)
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joel Bauer, Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 14-0377
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Ventral Incisional Hernia
Keywords: hernia repair; ventral incisional hernia; biologic mesh; hernia graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hernia graft/mesh: Hernia repair patients implanted with biologic hernia graft during surgery
  Interventions: Device: Hernia graft/mesh

INTERVENTIONS:
Device: Hernia graft/mesh — observational group
  Other Names: Cook Biodesign hernia graft

SUMMARY:
The purpose of this study is to evaluate the efficacy of the Cook Biodesign mesh for the repair of complex ventral incisional hernias. Using materials to reinforce tissue defects is indicated as standard of care for this type of surgery. The Cook Biodesign mesh is currently FDA-approved for implantation to reinforce soft tissues where weakness exists, but the investigators would like to collect additional follow-up information to continue to assess the durability of the repair after placement of the hernia mesh. This follow-up would include the collection of information about complications such as infections and seromas (collections of fluid around the surgery site), as well as hernia recurrence and quality of life questionnaires. Patients who qualify to take part in this study have been diagnosed with a ventral incisional hernia and will have been scheduled for a surgical hernia repair. This surgery will be an "open" surgical procedure and reinforcing your tissue with material is indicated for this type of hernia repair.

DETAILED DESCRIPTION:
Prior to their scheduled surgery, the patient will be consented and will complete a brief quality of life survey. They will also be asked some questions about their medical history that pertain to the study, such as current/ past abdominal infections and surgeries, history of the hernia, comorbidities, etc.

During the surgery, some key data points will be recorded by the research coordinator, such as time of surgery, type of case, size of mesh used, size of the hernia defect, technique used, type of sutures used, etc. The mesh will be placed either retrorectus or intraperitoneally, after the component separation is complete. The mesh will not be used as a "bridge," and the fascial layers will be closed completely.

The research staff may photograph the repair of an enrolled patient's hernia during their treatment and will supply a copy of the photograph to Cook Medical, Inc. if the sponsor's review is requested. Any photograph taken for research purposes will be kept in a password-protected, encrypted database separate from any patient identifying information.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a ventral incisional hernia repair with mesh
* Age range between 18 and 80 years old

Exclusion Criteria:

* Patients currently enrolled in a clinical trial.
* Patients with a BMI over 40
* Patients in whom the fascial layers cannot be closed or in whom "bridging" would be used
* Patients with a current abdominal abscess or infection
* Patients with healing disorders
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study team will screen the office schedules of the investigators for patients presenting for open bowel resection at the Mount Sinai Medical Center. Patients who meet the eligibility criteria will be asked if they are interested in volunteering to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Hernia Recurrence | up to 2 years
  Assessment of efficacy of the device and repair

SECONDARY OUTCOMES:
Infections | up to 2 years
  Infections related to the surgical site or implantation of the device
Seromas | up to 2 years
Rehospitalization | up to 2 years
Re-operation | up to 2 years
Mesh Removal | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joel J Bauer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States